CLINICAL TRIAL: NCT05891600
Title: Adherence and Clinical Outcomes in Patients With e-Device for Etanercept Administration in Rheumatoid Arthritis Patients: Real Word Evidence in a Colombian Institution.
Brief Title: A Study to Learn About the Adherence and Clinical Outcomes in Colombian Patients With an E-Device for Etanercept Administration in Rheumatoid Arthritis
Status: Terminated | Type: Observational
Why Stopped: The study was terminated following a comprehensive review of the collected data and an assessment of the study's completeness. This decision was made to maintain scientific standards and ethical conduct, and to prevent potentially inaccurate results
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1801421; NCT05891600 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-05-26; First posted 2023-06-07 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Observational study
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

GROUPS / COHORTS (1):
- Rheumatoid arthritis patients in Colombia
  Interventions: Drug: Etaneracept Smartclic

INTERVENTIONS:
Drug: Etaneracept Smartclic — The SmartClic® autoinjector is a reusable, electromechanical, and single-patient device for the administration of subcutaneously administered biologics.

SUMMARY:
This is a descriptive, ambispective, and single-site study in Colombia, which is designed to evaluate the adherence, persistence, and clinical outcomes (defined as the patient's disease activity and functional status) of RA patients within 40 weeks after the patient administered the first injection of the etanercept medication through the Smartclic® device. The study data seeks from medical records containing the Smartclic device injection log and pharmacy claims database available from an institution specialized in rheumatological care. The study will only include records of patients treated or starting treatment with etanercept and whose indicated autoinjection device has been Smartclic.

DETAILED DESCRIPTION:
Non-interventional study: The clinical records of eligible patients will be identified by the rheumatologist from the patients who attended the rheumatologist visit or institutional training sessions according to the standard of care. Patients have been prescribed etanercept according to the standard of care, and Smartclic has been indicated as an administration method.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.
* Patients aged ≥18 years with an established diagnosis of rheumatoid arthritis according to EULAR-ACR criteria recorded in medical record.
* Patients who are on etanercept treatment and are being switched to Smartclic, or new etanercept patients that have been prescribed Smartclic® device (either in combination with a conventional synthetic DMARD or in monotherapy).
* Medical records and pharmacy claims database of the IPS available after the index date for a period of 40 weeks.

Exclusion Criteria:

- Any serious ongoing infections, pregnancy, or other social or medical conditions that are anticipated in the investigator's judgment to lead to discontinuation of etanercept administration with the device during the 40 weeks of data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study data will be collected from medical records containing the Smartclic device injection log and pharmacy claims database available from a rheumatologist institution. The study will only include clinical records of patients who received treatment with etanercept and meet the selection criteria.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-06-06 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Adherence (Pharmacy claims source) | Baseline through week 40
  The percentage of patients with Percentage of days covered (PDC) ≥ 80%
Change From Baseline in Disease Activity Score Based on 28-joints Count with ESR (DAS28-ESR) at 40 week | Baseline, Week 40
Change From Baseline in Functional status Based on Multidimensional Health Assessment Questionnaire (MDHAQ) at 40 week | Baseline, Weeks 40

SECONDARY OUTCOMES:
Persistence | Week 40
  Number of days to discontinuation from the index date (date that the patient administered the first injection of the etanercept medication through the Smartclic device)
Adherence from Smartclic® injection log | Week 40
  Percentage of patients with administration ≥ 80% based on the injection log of the e-Device

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Biomab Ips S.A.S., Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1801421